CLINICAL TRIAL: NCT05779020
Title: A Blind Randomized Clinical Trial, With Active Controls, to Evaluate the Immunogenicity and Safety of the Quadrivalent Influenza Vaccine (Split Virion, Inactivated) From Instituto Butantan, in Infants and Children Aged 6 to 35 Months.
Brief Title: Immunogenicity and Safety of Butantan Quadrivalent Influenza Vaccine (Split Virion, Inactivated) in Infants and Children .
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Fundação Butantan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLQ-02-IB
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Influenza, Human
Keywords: Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QIV-IB/dose 0.25ml (Experimental): Butantan Quadrivalent Influenza Vaccine (split virion, inactivated)/dose 0.25ml
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated)
- QIV-IB/dose 0.50ml (Experimental): Butantan Quadrivalent Influenza Vaccine (split virion, inactivated)/dose 0.50ml
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated)
- TIVV-IB (Active Comparator): Butantan Trivalent Influenza Vaccine (split virion, inactivated)/dose 0.25ml containing Influenza B virus - Victoria lineage
  Interventions: Biological: Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Victoria lineage
- TIVY-IB (Active Comparator): Butantan Trivalent Influenza Vaccine (split virion, inactivated)/dose 0.25ml containing Influenza B virus - Yamagata lineage
  Interventions: Biological: Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Yamagata lineage

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) — Quadrivalent Influenza Vaccine (split virion, inactivated) from Instituto Butantan (dose 0.25ml and 0.50ml)
  Arms: QIV-IB/dose 0.25ml; QIV-IB/dose 0.50ml
Biological: Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Victoria lineage — Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Victoria lineage/dose 0.50ml
  Arms: TIVV-IB
Biological: Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Yamagata lineage — Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Yamagata lineage/dose 0.25ml
  Arms: TIVY-IB

SUMMARY:
This is a Phase III Randomized Clinical Trial, blind, multicenter, with active controls, to evaluate the immunogenicity and safety of the Quadrivalent Influenza Vaccine (split virion, inactivated) from Instituto Butantan, in two dose scheme (0.25ml and 0.50ml), in infants and children under 3 years of age.

DETAILED DESCRIPTION:
The study will be carried out in multiple sites in Brazil, using a community-based recruitment strategy.

The study interventions are the Butantan Quadrivalent Influenza Vaccine (split virion, inactivated) in two dose scheme (QIV-IB/0.25ml and QIV-IB/0.50ml) and the active controls Butantan Trivalent Influenza Vaccine (split virion, inactivated) containing Influenza B virus - Victoria or Yamagata lineage (TIVV-IB and TIVY-IB), in a ratio 1:1:1:1.

The study population is healthy infants and children aged 6 to 35 months and all participants will be followed up 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infant and child of either sex aged between 6 and 35 months on the day of the first study vaccination.
2. Born at term (≥ 37 weeks of gestational age) and birth weight ≥ 2.5 kg.
3. Parents/legal guardians of the infant or child able and willing to attend all scheduled visits and comply with all study procedures, including blood draws.
4. Parents/legal guardians of the infant or child have provided informed consent.

Exclusion Criteria:

1. Having received any influenza vaccine from the current season and/or 6 months before the first study vaccination.
2. History of allergy to egg, chicken proteins, or other components of the influenza vaccine.
3. History of serious adverse reaction to any influenza vaccine.
4. Have any clinically significant condition or situation that, in the Investigator's opinion, would interfere with study evaluations or participation.
5. History of Guillain-Barré or other demyelinating diseases.
6. History of neurological disease and/or clinically significant developmental delay (at the discretion of the Investigator), or seizure (except for an isolated febrile seizure episode).
7. Having received immune globulin, blood, or any blood product 3 months before the planned date of the first study vaccination or planned administration during the study period.
8. Any confirmed or suspected immunosuppressive condition, congenital or acquired immunodeficiency (including human immunodeficiency virus - HIV) based on medical history and physical examination.
9. Immediate personal or family history of congenital immunodeficiency.
10. Having received or are using radiation therapy, chemotherapy, immunosuppressive drugs, or other immunomodulatory drugs within three months before the planned date of the first study vaccination or planned use during the study.
11. Be a solid organ or bone marrow/stem cell transplant recipient.
12. Thrombocytopenia, bleeding disorder, use of anticoagulants, or any condition that contraindicates intramuscular injection.
13. Significant chronic disease (cancer, autoimmune disease, diabetes mellitus, acute or progressive liver disease, acute or progressive kidney disease, severe heart or lung disease) or which in the Investigator's opinion poses a risk to the health of the infant or child participating in the study or which may interfere with the conduct or conclusion of the study.
14. History of seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
15. Major surgery or surgery using general anesthesia planned to occur during the period between the first vaccination and 28 days after full vaccination in the study.
16. Any condition that, in the opinion of the Investigator, may interfere with the conduct or completion of the study (such as travelling or planned moving of residence, among others).
17. Participation in another clinical trial involving another experimental or unregistered product 1 year before the planned date of the study's first vaccination, or plans to entering a clinical trial during the study.
18. Infant and institutionalized child.
19. Be related to the Investigator, research site staff member, or employee directly involved in the study.

Postponement Criteria:

1. Have received any vaccine (including routine childhood vaccines) within 28 days of the first study vaccination (delay until the 28-day deadline from the date of the last vaccination).
2. Moderate or severe (as judged by the Investigator) acute illness/infection or febrile illness (temperature ≥ 37.8°C) 48 hours before the planned date of the first study vaccination.
3. Acute respiratory illness within 14 days preceding the planned date of the first study vaccination.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1373 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Ratio of Geometric Mean Titers (rGMT) of antibodies induced by QIV-IB/0.25ml compared to those induced by TIVV-IB and TIVY-IB, for each strain, in infants and children from 6 to 35 months of age. | 28 days after last vaccination
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.
Ratio of Geometric Mean Titers (rGMT) of antibodies induced by QIV-IB/0.50ml compared to those induced by TIVV-IB and TIVY-IB, for each strain, in infants and children from 6 to 35 months of age. | 28 days after last vaccination
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.
Ratio of Geometric Mean Titers (rGMT) of antibodies induced by QIV-IB/0.25ml compared to those induced by TIV that does not contain the B strain, for B lineage Victoria and Yamagata, in infants and children aged 6 to 35 months age. | 28 days after last vaccination
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.
Ratio of Geometric Mean Titers (rGMT) of antibodies induced by QIV-IB/0.50ml compared to those induced by TIV that does not contain the B strain, for B lineage Victoria and Yamagata, in infants and children aged 6 to 35 months age. | 28 days after last vaccination
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.

SECONDARY OUTCOMES:
Ratio of Geometric Mean Titers (rGMT) of antibodies induced by QIV-IB/0.50ml compared to those induced by QIV-IB/0.25ml, for each strain, in infants and children from 6 to 35 months of age. | 28 days after last vaccination
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.
Percentage of Participants With Seroconversion (Seroconversion Rate - SCR) to Influenza Vaccine Antigens. | At Days 0 and 28/56
  SCR is defined as the percentage of subjects with either a prevaccination HAI titer < 1:10 and a postvaccination HI titer ≥ 1:40, or a prevaccination HI titer ≥ 1:10 and a ≥ 4-fold increase in postvaccination HI titer.
Percentage of Participants achieving seroprotection (Seroprotection Rate - SPR) to Influenza Vaccine Antigens. | At Days 0 and 28/56
  Seroprotection Rate is defined as the percentage of subjects with HAI titer ≥1:40
Pre- and post-vaccination Geometric Mean Titers (GMT) induced by QIV-IB/0.25ml, QIV-IB/0.50ml, TIVV-IB e TIVY-IB, for each strain, in infants and children from 6 to 35 months of age. | At Days 0 and 28/56
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.
Ratio of Pre- and post-vaccination Geometric Mean Titers (rGMT) induced by QIV-IB/0.25ml, QIV-IB/0.50ml, TIVV-IB e TIVY-IB, for each strain, in infants and children from 6 to 35 months of age. | At Days 0 and 28/56
  Immunogenicity outcomes assessed in serum samples by hemagglutination inhibition (HAI) assay.
Solicited local Site or Systemic Reactions After each Injection | Day 0 up to Day 7 post-injection
  Percentage of subjects with Solicited local Site or Systemic Reactions After each Injection
Related Unsolicited Adverse Events | 28 days after last vaccination
  Percentage of subjects with Related Unsolicited Adverse Events
Serious Adverse Events (SAE) and adverse events of special interest (AESI) | Entire study participant's follow-up period (6 months after the last vaccination)
  Percentage of subjects with Serious Adverse Events (SAE) and adverse events of special interest (AESI)

CONTACTS AND LOCATIONS:
Locations (10):
- Brazil (10):
  - Instituto Auto Imune de Pesquisa e Educação Continuada - Real Hospital Português de Beneficência em Pernambuco (Site REC01), Recife, Pernambuco
  - Centro Oncológico de Roraima - CECOR (Site BVB-01), Boa Vista, Roraima
  - Centro de Pesquisas Clínicas da Universidade Federal de Sergipe (Site AJU01), Laranjeiras, Sergipe
  - Hospital das Clínicas da Faculdade de Medicina Ribeirão Preto - USP (Site RAO 04), Ribeirão Preto, São Paulo
  - Centro de Pesquisa Clínica S (Site RAO03), Serrana, São Paulo
  - CPMC Pesquisa Clínica - Clinica De Alergia Martti Antila Sorocaba, Sorocaba, São Paulo
  - A2Z Clinical Centro Avançado de Pesquisa Clínica Ltda.(Site 001), Valinhos, São Paulo
  - CPQuali Pesquisa Clínica Ltda (Site 002), São Paulo
  - Instituto de Pesquisa PENSI (Site SAO09), São Paulo
  - Centro de Pesquisa Clínica do Instituto da Criança - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (Site SAO08), São Paulo

IPD SHARING:
Plan to Share IPD: No